CLINICAL TRIAL: NCT04835389
Title: A Phase 1 Study Evaluating the Safety and Preliminary Efficacy of AlloGen® Liquid Intra-articular Injection for Knee Osteoarthritis
Brief Title: Study of AlloGen® Liquid Intra-articular Injection for Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: VIVEX Biologics, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-2021-001
Record Dates: First submitted 2020-12-11; First posted 2021-04-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; biologic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-Controlled, Double-Blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects and investigators (including outcomes assessment) will be blinded to the treatment arm that is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AlloGen Liquid (Experimental): A single-dose, intra-articular (IA) injection of 2.0 mL of AlloGen Liquid administered to the affected knee.
  Interventions: Biological: AlloGen Liquid
- Saline (Placebo Comparator): A single-dose, intra-articular (IA) injection of 2.0 mL of saline administered to the affected knee.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AlloGen Liquid — Amniotic fluid
  Arms: AlloGen Liquid
Drug: Placebo — 0.9% normal saline
  Arms: Saline

SUMMARY:
A randomized, double-blind, placebo-controlled trial comparing a single intra-articular injection of 2.0 mL AlloGen vs 2.0 mL sterile saline. Patients will be evaluated at baseline, 1 week, 6 weeks, 12 weeks, and 26 weeks.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled trial comparing a single intra-articular 2.0 mL injection of either AlloGen or sterile saline. Patients will be evaluated at baseline, 1 week, 6 weeks, 12 weeks, and 26 weeks. The patient will remain blinded to his or her treatment throughout the study duration. The investigator/assessor will also remain blinded throughout the treatment period. Only the individual(s) preparing the injection will not be blinded. Black tape over the injection syringe will mask the study treatment.

Up to 30 adult patients with osteoarthritis of one knee that has failed to adequately respond to conservative non-pharmacologic therapy and simple analgesics, e.g., acetaminophen, will be enrolled at up to 5 sites in the US. The first 6 subjects will be staggered to evaluate any significant toxicity. Any adverse event data collected will be reviewed by the Data Safety Monitoring Board (DSMB) prior to treating the subsequent subject. Cumulative safety data from these 6 subjects will be reviewed by the DSMB.

ELIGIBILITY:
Inclusion Criteria:

* Subject has both clinical and radiographic findings consistent with osteoarthritis of the knee:

  1. Subject has clinical findings including (but not limited to) tenderness to palpation, swelling/effusion, stiffness, chronic limited range of motion.
  2. Subject has a diagnosis of knee osteoarthritis (OA) defined as Grade 2 to 3 using the Kellgren-Lawrence grading scale.
* Failed conservative care over the past 3 months of at least 2 conservative treatments including oral pain medication [analgesics, steroids and/or non-steroidal anti-inflammatory drugs (NSAIDs)] and structured physical therapy or exercise program prescribed by physical therapist, chiropractor provider or physician specifically for the treatment of knee osteoarthritis.
* Subject has a BMI less than 40 kg/m2
* Subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study.
* Subject must have a VAS pain score of 4 or greater on a 100-mm scale.
* All subjects of reproductive age or capacity must use adequate contraception (abstinence, surgically sterilized, postmenopausal, or consistently use an effective contraception method) during the study.
* Subject agrees not to take additional knee symptom-modifying drugs (e.g., glucosamine, collagen, hyaluronic acid) during the study without reporting the use to the study team.

Exclusion Criteria:

* Subject has a diagnosis of knee osteoarthritis (OA) defined as Grade 4 on the Kellgren-Lawrence grading scale.
* Subject has active infection at the injection site.
* Subject has symptomatic OA of the contralateral knee or of either hip (VAS≥40) that is not responsive to acetaminophen (Tylenol®) and/or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs, e.g. Ibuprofen) and requires other therapy.
* Subject has rheumatoid arthritis, psoriatic arthritis, or has been diagnosed with any other disorders that is the primary source of their knee pain, including but not limited to:

osteonecrosis, radiculopathy, bursitis, tendinitis, tumor, cancer.

* Subject has documented history of gout or pseudo-gout.
* Subject has a known allergy to local anesthetics.
* Subject has autoimmune disease or a known history of having Acquired Immunodeficiency Syndromes (AIDS) or Human Immunodeficiency Virus (HIV).
* Subject has diagnosis of hematologic, renal, hepatic, or coagulation abnormalities based on medical history and laboratory results.
* Subject has received any of the following to the target knee:

  1. Intra-articular hyaluronic acid (HA) injection within 12 weeks prior to screening;
  2. Steroid or platelet rich plasma (PRP) injection within 12 weeks prior to screening;
  3. Has had or is planning to have major surgery in the target knee within 26 weeks of treatment; or
  4. History of unicondylar or total knee arthroplasty.
* Subject is currently participating in another clinical trial or has used an investigational drug, device or biologic within 12 weeks prior to treatment.
* Subject has a history of immunosuppressive use or chemotherapy in the last 12 months.
* Subject has had prior radiation to the index knee.
* Subject is currently taking anticoagulant therapy (excluding Plavix or Aspirin).
* Subject is breast feeding or pregnant or plans to become pregnant within 12 weeks of treatment.
* Subject has any significant medical condition that, in the opinion of the Investigator, would increase the chances of an adverse event and/or would interfere with protocol evaluation and participation.
* Subject is a worker's compensation patient.
* Subject has taken pain medication <48 hours prior to the injection or has received pain medicine other than acetaminophen and/or NSAIDs for conditions unrelated to OA of the index knee.
* Subject has a history of alcohol or substance abuse.
* Physical or IA injection exclusion criteria include:

  1. Frank mechanical symptoms such as locking, intermittent block to range of motion, or loose body sensations (meniscal displacement or IA loose body),
  2. Knee surgery on index knee within 12 months or on contralateral knee within 6 months, and/or
  3. Acute injury to the knee within 3 months.
* Subject has uncontrolled, unstable diabetes mellitus with HbA1C =/>8%.
* History within preceding 5 years of solid organ or hematologic transplantation or diagnosis of non-basal cell malignancy.
* History within the preceding 6 months of septic arthritis in the affected knee or sepsis/bacteremia.
* History within the preceding 3 months of infection requiring antibiotic treatment .

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of intra-articular (IA) administration of AlloGen Liquid in the target knee | Baseline to 12 weeks
  The incidence of related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events

SECONDARY OUTCOMES:
Evaluate preliminary efficacy of the injection by assessing pain subscale scores | Baseline, 6, 12 and 26 weeks
  Composite change from baseline in WOMAC-A (pain subscale) scores
Evaluate preliminary efficacy of the injection by assessing function subscale scores | Baseline, 6, 12 and 26 weeks
  Composite change from baseline in WOMAC-C (function subscale) score
Evaluate preliminary efficacy of the injection by assessing pain | Baseline, 6, 12 and 26 weeks
  Change from baseline in WOMAC-A scores
Evaluate preliminary efficacy of the injection by assessing function | Baseline, 6, 12 and 26 weeks
  Change from baseline in WOMAC-C score
Evaluate preliminary efficacy of the injection by Visual Analog Scale | Baseline, 6, 12 and 26 weeks
  Change from baseline in Visual Analog Scale (VAS)
Evaluate preliminary efficacy of the injection by assessing total WOMAC | Baseline, 6, 12 and 26 weeks
  Change from baseline in total WOMAC score
Evaluate the safety of intra-articular (IA) administration of AlloGen Liquid in the target knee | 26 Weeks
  Incidence of related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events at 26 weeks
Evaluate preliminary efficacy of the injection by assessing Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 6, 12 and 26 weeks
  Change from baseline in PROMIS pain interference and physical function scores
Evaluate preliminary efficacy of the injection by assessing total SF-12 score | Baseline, 6, 12 and 26 weeks
  Change from baseline in total SF-12 score
Evaluate preliminary efficacy of the injection by assessing total KOOS score | Baseline, 6, 12 and 26 weeks
  Change from baseline in total KOOS score

CONTACTS AND LOCATIONS:
Overall Officials: Brian Cole, MD, Principal Investigator — Brian Cole MD

IPD SHARING:
Plan to Share IPD: No